CLINICAL TRIAL: NCT01938235
Title: Exenatide for Myocardial Protection During Reperfusion Study: A Double-blind, Placebo-controlled Trial
Brief Title: Exenatide for Myocardial Protection During Reperfusion Study
Acronym: EMPRES
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Vladimír Džavík, Director, Research and Innovation in Interventional Cardiology and Cardiac Intensive Care, Division of Cardiology, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB001-001; 9427-D0416-21C (Other: Health Canada)
Record Dates: First submitted 2013-08-29; First posted 2013-09-10 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Percutaneous coronary intervention; Reperfusion injury; Exenatide; Magnetic resonance imaging
MeSH Terms: conditions — Myocardial Infarction; Reperfusion Injury | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Experimental): o Exenatide at a dose of 1.5 µg IV over 30 min followed by 1.2 µg/hr IV for 1.5 h (Rate1), followed by 1.9 µg/hr IV* for 22 h (Rate 2)
  *Once the creatinine clearance is available, if the value is <60 mL/min, the rate at 2 hours will be maintained at Rate 1 for the duration of the infusion. If the value becomes available after the 2-hour point, and the rate has already been changed to Rate 2, the infusion will be titrated back down to Rate 1 if the creatinine clearance is <60 mL/min.
  If the creatinine clearance is <30 mL/min, the infusion will be discontinued and the patient will otherwise continue with all study procedures.
  A bolus administration of study medication is initiated preferably prior to reperfusion, or, if not possible, up to 30 minutes after the start of reperfusion to avoid delays in door-to-door balloon times.
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): o Placebo bolus over 30 min followed by placebo infusion at 'Rate 1' for 1.5 h, followed by 'Rate 2' for 22 hours*.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — Intravenous bolus and 24-hour infusion of exenatide
  Other Names: Byetta
  Arms: Exenatide
Drug: Placebo — Intravenous bolus and 24-hour infusion of placebo
  Arms: Placebo

SUMMARY:
This study aims to assess the effect of exenatide on myocardial injury in patients undergoing emergent percutaneous coronary intervention (PCI) for ST segment elevation myocardial infarction or heart attack (STEMI).

DETAILED DESCRIPTION:
This is a Phase II randomized, double-blind, placebo-controlled study of patients with STEMI. Those who agree to participate will be immediately randomized to one of two groups: a 24-h infusion of exenatide; or a 24 h infusion of placebo. We will assess the ability of exenatide to reduce ischemic injury. This study will serve as safety evaluation study as well as a pilot for a larger multicentre trial powered for clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Admission for primary PCI for STEMI, with enrollment within 12 hours of onset of symptoms. STEMI will be defined as typical ECG changes (ST segment elevation ≥1mm in 2 or more limb leads, or ≥2mm in 2 or more precordial leads, or new onset LBBB) associated with acute chest pain or an elevation of cardiac enzymes.
* Antegrade TIMI 0 or 1 prior to PCI in the infarct-related artery
* Age ≥18 years

Exclusion Criteria:

* Symptomatic hypoglycemia (serum glucose <3.3 µmol/L; 60 mg/dl)
* Diabetes mellitus requiring insulin therapy
* Diabetic ketoacidosis
* Coronary anatomy warranting emergent coronary artery bypass graft surgery
* Mechanical complication of STEMI (ventricular septal rupture, free wall rupture, acute severe mitral regurgitation)
* Need for hemodialysis
* Malignancy, HIV, or central nervous system disorder
* Cardiopulmonary resuscitation >15 min and compromised level of consciousness.
* Cardiogenic shock
* Current participation in any research study involving investigational drugs or devices
* Inability to give informed consent
* Inability to safely undergo cMRI (presence of cardiac pacemaker, implanted cardiac defibrillator, aneurysm clips, carotid artery vascular clamp, neurostimulator, implanted drug infusion device, bone growth/fusion stimulator, cochlear, otologic, or ear implant, severe claustrophobia)
* Women of childbearing potential who are known to be pregnant or lactating or who have a positive pregnancy test on admission
* History of pancreatitis
* Known end stage renal failure or known eGFR <30 mL/min
* Currently taking exenatide (Byetta, Bydureon), liraglutide (Victoza), or any other GLP-1 agonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-07 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Ratio of final infarct size at 3 months over area at risk at 72 hours post randomization (using cMRI) | 3 months

SECONDARY OUTCOMES:
Left ventricular global and regional LV systolic ejection fraction | 72 hours
Left ventricular global and regional LV systolic ejection fraction | 3 months
Left ventricular volume | 72 hours
Left ventricular volume | 3 months
Infarct size/area of risk (measured by cMRI) | 3 months
Myocardial enzyme levels (troponin I and CK-MB) | 24 hours
ST segment elevation resolution (measured by ECG) | 1 hour
ST segment elevation resolution (measured by ECG) | 24 hours
ST segment elevation resolution (measured by ECG) | 72 hours
ST segment elevation resolution (measured by ECG) | 3 months
Angiographic myocardial blush score | At the time of the PCI procedure
Serum glucose concentration | Baseline
Serum glucose concentration | 8 hours
Serum glucose concentration | 16 hours
Serum glucose concentration | 24 hours
Serum glucose concentration | 72 hours
Inflammatory marker levels (interleukin-6, interleukin-10, TNF-alpha) | 24 hours
NT-proBNP blood levels | 24 hours
Death | 3 months
Myocardial infarction (heart attack) | 3 months
Measure of extent of heart failure (NYHA classification) | 72 hours
Measure of extent of heart failure (NYHA classification) | 3 months
Major adverse cardiac events (defined as a combined outcome of death, recurrent myocardial infarction, stroke, and unplanned repeat revascularization) | 6 months
Death | 6 months
Recurrent myocardial infarction (heart attack) | 6 months
Stroke | 6 months
Unplanned repeat revascularization | 6 months
Development of heart failure | 6 months
Cardiogenic shock | During index hospitalization (up to 6 months)
Blood glucose < 3.0 mmol/L | During index hospitalization (up to 6 months)
Hypotension (defined as SBP <90 mmHg) | During index hospitalization (up to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, MD, Study Chair — University Health Network, Toronto
Locations (10):
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Hamilton Health Sciences - General Site, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Quebec (Hopital Laval), Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided